CLINICAL TRIAL: NCT05689606
Title: The Relationship of Cortical Excitability, Cognitive Functions, and Peripheral Signaling Molecules Following Acute Exercise
Brief Title: Cortical Excitability, Cognitive Functions, and Peripheral Signaling Molecules
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Collaborators: Gazi University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 12091985
Record Dates: First submitted 2022-10-10; First posted 2023-01-19 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: HIIT; TMS; BDNF; Cathepsin B; cognitive performance
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise group (Experimental): The exercise group performs acute high-intensity interval training.
  Interventions: Behavioral: Exercise
- Control group (No Intervention): The Control group includes the same participants. In this session, they do not exercise, and they watch a nature documentary.

INTERVENTIONS:
Behavioral: Exercise — Exercise includes acute high-intensity interval training.
  Arms: Exercise group

SUMMARY:
It is widely known that exercise creates structural and functional changes in the brain. Synaptic plasticity develops through exercise, thus improving brain functions. It is suggested that skeletal muscle contraction and peripheral signal molecules secreted from various tissues, especially skeletal muscle, contribute to exercise's effect on the brain's structure and function. These signals synthesized and released from skeletal muscle are called myokines. Brain-derived neurotrophic factor (BDNF) and Cathepsin B are two of these myokines, which have been reported to cross the blood-brain barrier following secretion in the periphery and affect the structure and functions of the brain. Transcranial magnetic stimulation (TMS) allows to evaluate the synaptic plasticity responses of the motor cortex to exercise, while cognitive function responses are evaluated via cognitive tests. Additionally, exercise type and intensity influence the responses of cortical excitability and cognitive function. This research proposal aims to investigate how acute high-intensity intermittent exercise (HIIT) changes primary motor cortex (M1) excitability, M1-related cognitive functions, and peripheral BDNF and Cathepsin B levels in healthy sedentary adults and to investigate the relationship between these neurophysiological parameters. All parameters will be measured before and after the acute exercise. M1 excitability will be evaluated through resting motor threshold, short interval intracortical inhibition, and input-output curve measurements. Cognitive functions will be evaluated through mental rotation and working memory tasks, and peripheral signal responses will be measured by serum levels of BDNF and Cathepsin B. Our hypotheses are: 1) Acute HIIT will increase peripheral BDNF and CTSB level, cortical excitability, and M1-specific cognitive function performance. 2) M1 excitability, cognitive function performance, and peripheral BDNF and CTSB increase will be related following exercise. Our findings will have the potential to be a guide for the integration of exercise into daily life and will provide cortical and peripheral data on the neurophysiological basis of the relationship between exercise and cognition.

DETAILED DESCRIPTION:
Participants Twenty-eight healthy young adults (female|male:14|14) aged 20-30 years will have participated in the study.

Participants will be at least undergraduate students, right-handed dominant, exercising <150 minutes per week in the last six months. Before the experiment, the participants will be evaluated for their background, family history, and whether they have any health complaints that prevent them from exercising.

With the adult transcranial magnetic stimulation safety screening questionnaire, participants in the risk group for brain stimulation, those with intracranial implants and contraindications, and those with a history of any psychiatric or neurological disease, seizures, any serious medical condition, or pregnancy will be excluded. The hand preference questionnaire will evaluate hand preference, and physical activity status will be evaluated by the short version of the international physical activity questionnaire. The cardiorespiratory fitness will be assessed with the graded maximal exercise stress test. The N-back test is a continuous performance test used to assess working memory capacity. The mental rotation test will evaluate the mental rotation score. The research team designed both tests.

Transcranial magnetic stimulation will be used to assess corticomotor excitability. Resting Motor Threshold (RMT), Short Interval Intracortical Inhibition (SICI), and input-output curve measurements will be performed on all participants in our study for the TMS study.

BDNF and CTSB measurements of the participants will be made both at baseline and following the acute exercise.

HIIT exercise lasting 23 minutes will be performed on the bicycle ergometer. Participants will make 3 visits to the laboratory. First session: Cardiorespiratory fitness assessment, all questionnaires. Second session: TMS analyses, cognitive assessments, HIIT, myokine assessments Third session: TMS analyses, cognitive assessments, control (watching a nature documentary).

The second and third sessions will be performed by cross-over design. Data analysis will be performed with two-way repeated ANOVA to determine the effect of within-group factors (control and HIIT) and time (PRE and POST) on corticospinal excitability and other parameters. When the effect size was calculated as ɳp2 >0.26, the sample size was calculated a priori as n = 22. Considering possible data losses, the number of participants was determined as 28.

ELIGIBILITY:
Inclusion Criteria:

* Being right-handed
* Aged between 20 and 30 years
* Being sedentary

Exclusion Criteria:

* having intracranial implants
* history of psychiatric or neurological disease, seizure, any serious medical condition or pregnancy

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Resting motor threshold | Change from Baseline resting motor threshold immediately following acute exercise
  The amount of transcranial magnetic stimulation machine output necessary to produce a motor-evoked potential that exceeds a defined peak-to-peak amplitude. Lower scores mean a better outcome.
Short interval intracortical inhibition | Change from Baseline short interval intracortical inhibition immediately following acute exercise
  The relative amplitude reduction of motor evoked potentials by subthreshold conditioning stimuli.
Input output curve | Change from Baseline input output curve immediately following acute exercise
  The input-output curve is a sigmoid-shaped relation between the MEP amplitude at incremented TMS intensities. Higher scores mean a better outcome.
Working memory | Change from Baseline working memory score immediately following acute exercise
  The small amount of information that can be held in mind and used in the execution of cognitive tasks. Higher scores mean a better outcome.
Serum BDNF | Change from Baseline serum BDNF immediately following acute exercise
  Serum level of BDNF. Higher scores mean a better outcome.
Mental rotation | Change from Baseline mental rotation score immediately following acute exercise
  The ability to transform a mental representation of an object so as to accurately predict how the object would look from a different angle. Higher scores mean a better outcome.
Serum Cathepsin B | Change from Baseline serum Cathepsin B immediately following acute exercise
  Serum level of Cathepsin B. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No